CLINICAL TRIAL: NCT06648577
Title: 3D Ultrasound Myocardial Mechanical Wave Measurements in Primary Mitral Regurgitation
Brief Title: 3D Ultrasound Myocardial Mechanical Wave Measurements
Acronym: 3DUsMR
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP 240537; IDRCB (Other: 2024-A01637-40)
Record Dates: First submitted 2024-10-10; First posted 2024-10-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Chronic Primary Mitral Regurgitation
Keywords: Primary mitral regurgitation; High frame rate ultrasound imaging; CMR; Myocardial fibrosis
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Comprehensive 2D/3D echocardiography: This an observational non interventional study. All patients will have both comprehensive 2D/3D echocardiography (including MWV imaging) and cardiac CMR.
  Interventions: Procedure: Ultrasound imaging

INTERVENTIONS:
Procedure: Ultrasound imaging — The participants are scanned with an ultrasound scanner

SUMMARY:
Primary mitral regurgitation (MR) is a frequent disease that can ultimately lead to heart failure. Primary MR represents the second most prevalent cause of cardiac valve surgery in high income countries. Progressive myocardial fibrosis due to chronic volume overload is recognized as a pathophysiological substrate of altered LV function in primary MR. As fibrosis leads to increased myocardial stiffness, ultrasound mechanical wave propagation measurements within the myocardium could provide important clinical information. Natural mechanical wave velocity (MWV) imaging, using High-frame-rate (HFR) echocardiography has emerged as a promising tool to evaluate myocardial stiffness.

The objective is study is to evaluate the correlation between the LV myocardial stiffness (as assessed by 3D ultrasound myocardial MWV mapping) and myocardial interstitial fibrosis as measured using CMR (myocardial extracellular volume measure)

DETAILED DESCRIPTION:
After being informed about the study. All patients giving written informed consent will undergo in a routine practice:

1. echocardiography (2D/3D),
2. CMR imaging,
3. electrocardiogram 24 hours monitoring,
4. blood sampling including brain natriuretic peptide measurement,
5. symptom-limited combined exercise echocardiography and oxygen uptake measurements

ELIGIBILITY:
Inclusion Criteria:

* Severe primary MR patients (effective regurgitation orifice area ≥ 40mm²) with class I indication for surgery (symptoms and/or altered conventional parameters of LV function) (n=10 patients)
* Severe primary MR patients (effective regurgitation orifice area ≥ 40mm²) without class I indication of surgery (n=20 patients)
* Mild to moderate primary MR patients as defined by effective regurgitation orifice area ≥ 20mm² and < 40mm² (n=10 patients)

Exclusion Criteria:

* Permanent atrial fibrillation
* Acute primary severe MR
* Secondary MR
* Previous cardiac surgery of any kind
* Other severe left sided valvular disease
* Coronary artery disease
* Congenital cardiac disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include adult patients with chronic primary mitral regurgitation who have been referred to our tertiary cardiology center as part of their routine care. These are the typical patients with chronic primary mitral regurgitation whom we aim to better phenotype using the new 3D ultrasound mapping technology for MWV (mechanical wave velocity).
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2026-11-15 (Estimated); Study Completion 2027-11-14 (Estimated)

PRIMARY OUTCOMES:
To assess the correlation between left ventricular stiffness as assessed by 3D Mechanical wave velocity and myocardial fibrosis assessed with CMR (ECV measure). | baseline
  The speed of the mechanical wave in left ventricle will be measured (in m/s) using 3D high frame rate ultrasound imaging.
  Left ventricular interstitial fibrosis will be assessed by the measure of myocardial extracellular volume fraction (ECV, in %) by CMR.

SECONDARY OUTCOMES:
To assess the correlation between left ventricular stiffness as assessed by 3D Mechanical wave velocity and myocardial fibrosis assessed with CMR (T1 mapping) | baseline
  The speed of the mechanical wave in left ventricle will be measured (in m/s) using 3D high frame rate ultrasound imaging.
  Left ventricular fibrosis will be assessed from CMR by pre and post contrast T1 mapping (in milliseconds)
To assess the link between left ventricular stiffness as assessed by 3D Mechanical wave velocity and the 3 different clinical stages of chronic mitral regurgitation | baseline
  The speed of the mechanical wave in left ventricle will be measured (in m/s) using 3D high frame rate ultrasound imaging.
  The clinical stages of the patients are defined as follow:
  * Severe primary MR patients (effective regurgitation orifice area ≥ 40mm²) with class I indication for surgery (symptoms and/or altered LV function as defined by left ventricular ejection fraction ≤60% and/or left ventricular end systolic diameter ≥40mm) (n=10 patients)
  * Severe primary MR patients (effective regurgitation orifice area ≥ 40mm²) without class I indication of surgery (n=20 patients)
  * Mild to moderate primary MR patients as defined by effective regurgitation orifice area ≥ 20mm² and < 40mm² (n=10 patients)
To assess the correlation between left ventricular stiffness as assessed by 3D Mechanical wave velocity, left ventricular mass and global longitudinal strain | baseline
  The speed of the mechanical wave in left ventricle will be measured (in m/s) using 3D high frame rate ultrasound imaging.
  Left ventricular mass will be measured (in grammes /m²) using echocardiography and CMR Global longitudinal strain (in %) will be measured from echocardiography and CMR from apical 4, 2 and 3 chambers views.

OTHER OUTCOMES:
To assess the correlation between left ventricular stiffness as assessed by 3D Mechanical wave velocity and exercice capacity | 1 year
  The speed of the mechanical wave in left ventricle will be measured (in m/s) using 3D high frame rate ultrasound imaging.
  The exercise capacity will be measured thought symptom-limited combined exercise echocardiography and oxygen uptake measurements (in watts and using peak oxygen uptake expressed as mL/kg)
To assess the correlation between left ventricular stiffness as assessed by 3D Mechanical wave velocity and mitral regurgitation severity | 1 year
  The speed of the mechanical wave in left ventricle will be measured (in m/s) using 3D high frame rate ultrasound imaging.
  Mitral regurgitation severity will be assessed by echocardiography (effective regurgitation orifice area in mm² and regurgitation volume in mL) and using CMR (regurgitation orifice area, volume and regurgitation fraction).

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Pitié Salpêtrière hospital, Paris, Paris
  - Pitié- Salpêtrière hospital (AP-HP), Paris, Paris

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Salles S, Espeland T, Molares A, Aase SA, Hammer TA, Stoylen A, Aakhus S, Lovstakken L, Torp H. 3D Myocardial Mechanical Wave Measurements: Toward In Vivo 3D Myocardial Elasticity Mapping. JACC Cardiovasc Imaging. 2021 Aug;14(8):1495-1505. doi: 10.1016/j.jcmg.2020.05.037. Epub 2020 Aug 26. PMID 32861651